CLINICAL TRIAL: NCT00447005
Title: A Phase 1 Study Of AG-013736 (Axitinib) In Japanese Patients With Advanced Solid Tumors
Brief Title: Study Of AG-013736 (Axitinib) In Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4061022
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Carcinoma
Keywords: Safety; PK; Biomarker
MeSH Terms: conditions — Carcinoma | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open (Experimental)
  Interventions: Drug: Axitinib (AG-013736)

INTERVENTIONS:
Drug: Axitinib (AG-013736) — AG-013736 5mg twice daily [BID]

SUMMARY:
To evaluate the clinically recommended dose of AG-013736 (Axitinib) in Japanese patients by reviewing the safety of AG-013736 (Axitinib) following single and multiple dosing.

ELIGIBILITY:
Inclusion Criteria:

* Patients histologically or cytologically diagnosed with advanced malignant solid tumors
* Patients for whom standard therapies have not been effective, or for whom there are no suitable therapies

Exclusion Criteria:

* Central lung lesions involving major blood vessels
* Patients who have been treated with bevacizumab or other VEGFR inhibitor(s)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Kashiwa, Chiba, Japan

REFERENCES:
- [Derived] Mukohara T, Nakajima H, Mukai H, Nagai S, Itoh K, Umeyama Y, Hashimoto J, Minami H. Effect of axitinib (AG-013736) on fatigue, thyroid-stimulating hormone, and biomarkers: a phase I study in Japanese patients. Cancer Sci. 2010 Apr;101(4):963-8. doi: 10.1111/j.1349-7006.2009.01465.x. Epub 2009 Dec 9. PMID 20180805
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061022&StudyName=Study%20Of%20%20AG-013736%20%28Axitinib%29%20In%20Patients%20With%20Advanced%20Solid%20Tumors

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Six participants initially received a single dose of AG-013736 5 mg followed by 5 mg twice daily (BID) multiple dosing. They were monitored for dose limiting toxicity (DLT) up to multiple dosing Cycle 1. Since no more than 1 of the first 6 participants had a DLT, 6 additional participants initiated AG-013736 from multiple dosing per the protocol.
Groups:
- AG-013736: Single dose (first 6 participants only): Single AG-013736 5 mg was administered orally.
  Multiple dose (all participants): AG-013736 5 mg twice daily (BID) was administered orally in fed state, 12 hours apart at approximately the same time each day. AG-013736 dose was titrated or reduced based on the dose modification criteria: the available dose was 2, 3, 5, 7, or 10 mg at a time. One cycle length was 28 days and participants continued the study treatment until intolerable toxicity or disease progression occurred.
Period: Overall Study
Arm/Group | AG-013736
Started | 12
Completed | 0
Not Completed | 12
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 11

BASELINE CHARACTERISTICS:
Arm/Group | AG-013736
Number analyzed (Participants) | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 60.2 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants with any adverse events, adverse events graded as Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE) Grade 3 or higher, serious adverse events, and adverse events resulted in discontinuation.
Time Frame: Up to 795 days of treatment plus 28-days follow-up
Population: All subjects who received at least 1 dose of the study drug.
Measure: Number; unit: participants
Arm/Group | AG-013736
Number analyzed (Participants) | 12
participants
  Any adverse events | 12
  Any serious adverse events | 5
  Any Grade-3 or -4 adverse events | 7
  Any Grade-5 adverse events (= death) | 0
  Discontinuation due to adverse events | 1

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax): Single Dose
Time Frame: Single dose: predose, 0.5, 1, 2, 4, 6, 8, 12, 24, and 32 hours postdose
Population: Participants who received at least one study drug and completed pharmacokinetic blood sampling for at least one day (Pharmacokinetic Analysis Set). Only the first 6 participants were administered a single dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AG-013736
Number analyzed (Participants) | 6
ng/mL | 29.97 (9.97)

3. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax): Single Dose
Time Frame: Single dose: predose, 0.5, 1, 2, 4, 6, 8, 12, 24, and 32 hours postdose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | AG-013736
Number analyzed (Participants) | 6
hours | 4 [2 to 6]

4. Secondary Outcome: Area Under The Plasma Concentration-Time Curve From Time Zero to Time Infinity (AUCinf): Single Dose
Description: AUCinf is obtained from AUC (0 - t) plus AUC (t - infinity).
Time Frame: Single dose: predose, 0.5, 1, 2, 4, 6, 8, 12, 24, and 32 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | AG-013736
Number analyzed (Participants) | 6
ng*hr/mL | 210.3 (146.5)

5. Secondary Outcome: Terminal Phase Plasma Half-Life (t1/2): Single Dose
Description: t1/2 is the time measured for the plasma concentration to decrease by one half.
Time Frame: Single dose: predose, 0.5, 1, 2, 4, 6, 8, 12, 24, and 32 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | AG-013736
Number analyzed (Participants) | 6
hours | 4.8 (1.146)

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax): Multiple Dose
Time Frame: Multiple dose Cycle 1 Day 1 and 15: predose, 0.5, 1, 2, 4, 8 and 12 hours postdose
Population: Participants who received at least one study drug and completed pharmacokinetic blood sampling for at least one day (Pharmacokinetic Analysis Set); n= number of participants assessed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AG-013736
Number analyzed (Participants) | 12
ng/mL
  Cycle 1 Day 1 (n=12) | 23.85 (10.94)
  Cycle 1 Day 15 (n=11) | 32.14 (18.04)

7. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax): Multiple Dose
Time Frame: Multiple dose Cycle 1 Day 1 and 15: predose, 0.5, 1, 2, 4, 8 and 12 hours postdose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | AG-013736
Number analyzed (Participants) | 12
hours
  Cycle 1 Day 1 (n=12) | 3 [2 to 4]
  Cycle 1 Day 15 (n=11) | 4 [1 to 4]

8. Secondary Outcome: Area Under The Plasma Concentration-Time Curve Over Dosing Interval Tau (AUCtau): Multiple Dose
Description: Dosing Interval was 12 hours in this study.
Time Frame: Multiple dose Cycle 1 Day 1 and 15: predose, 0.5, 1, 2, 4, 8 and 12 hours postdose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | AG-013736
Number analyzed (Participants) | 12
ng*h/mL
  Cycle 1 Day 1 (n=12) | 137.3 (84.3)
  Cycle 1 Day 15 (n=11) | 187.8 (125.3)

9. Secondary Outcome: Accumulation Ratio for Cmax (Rac Cmax) and Accumulation Ratio for AUCtau (Rac AUCtau): Multiple Dose
Description: Rac Cmax is obtained from Cmax (Cycle 1, Day 15) divided by Cmax (Cycle 1, Day 1) Rac AUCtau is obtained from AUCtau (Cycle 1, Day 15) divided by AUCtau (Cycle 1, Day 1)
Time Frame: Multiple dose Cycle 1 Day 1 and 15: predose, 0.5, 1, 2, 4, 8 and 12 hours postdose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | AG-013736
Number analyzed (Participants) | 12
ratio
  Rac Cmax (n=11) | 1.449 (0.471)
  Rac AUCtau (n=11) | 1.541 (0.489)

10. Secondary Outcome: Percent Change From Baseline in Soluble Vascular Endothelial Growth Factor Receptor 2 and 3 (s-VEGFR2 and s-VEGFR3), Vascular Endothelial Growth Factor (VEGF), Soluble Stem Cell Factor Receptor (s-KIT)
Description: Percent change from baseline is obtained from (observed value minus baseline value) divided by baseline value multiplied by 100 in each parameter, i.e., VEGFR2, s-VEGFR3, s-KIT, and VEGF.
Time Frame: Prior to the initial dose (baseline), Day 1 of Cycle 2 and at the discontinuation
Population: Participants who received at least one study drug and completed pharmacodynamic blood sampling for at least one day (Pharmacodynamic Analysis Set); n= number of participants assessed.
Measure: Median (Full Range); unit: percent change
Arm/Group | AG-013736
Number analyzed (Participants) | 12
percent change
  s-VEGFR2: Cycle 2 Day 1 (n=12) | -41.73 [-53.2 to -10.1]
  s-VEGFR2: At discontinuation (n=11) | -40.57 [-53.0 to -8.4]
  s-VEGFR3: Cycle 2 Day 1 (n=12) | -52.50 [-93.7 to -15.6]
  s-VEGFR3: At discontinuation (n=11) | -65.48 [-81.2 to 39.4]
  s-KIT: Cycle 2 Day 1 (n=12) | -0.26 [-23.8 to 33.5]
  s-KIT: At discontinuation (n=11) | 4.66 [-31.2 to 12.9]
  VEGF: Cycle 2 Day 1 (n=12) | 266.92 [14.9 to 1030.4]
  VEGF: At discontinuation (n=11) | 43.48 [-15.5 to 423.1]

11. Secondary Outcome: The Numbers of Participants With Best Overall Response of Complete Response (CR), Partial Response (PR), Stable Disease (SD), and Progression of Disease (PD) According to the Response Evaluation Criteria in Solid Tumors (RECIST Version 1.0)
Description: CR was defined as the disappearance of all target and nontarget lesions and no appearance of new lesions. PR was defined as at least a 30% decrease in the sum of the longest diameters (SLD) of the targeted lesions. CR and PR had to be documented on 2 occasions separated by at least 4 weeks. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify as PD being demonstrated during the first 8 weeks. PD was defined as at least a 20% increase in the SLD of target lesions compared to the smallest SLD since the study treatment started.
Time Frame: Up to 795 days
Population: Participants with at least 1 target lesion according to RECIST and who received at least 1 dose of study drug (Anti-tumor Response Analysis Set).
Measure: Number; unit: participants
Arm/Group | AG-013736
Number analyzed (Participants) | 12
participants
  CR | 0
  PR | 0
  SD | 10
  PD | 2

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | AG-013736
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AG-013736 (N=12)
Cardiac tamponade (Cardiac disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 2
Liver abscess (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AG-013736 (N=12)
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 10
Dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Proctalgia (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 9
Toothache (Gastrointestinal disorders) | 2
Face oedema (General disorders) | 1
Fatigue (General disorders) | 10
Generalised oedema (General disorders) | 1
Pyrexia (General disorders) | 1
Thirst (General disorders) | 1
Herpes zoster (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Onychomycosis (Infections and infestations) | 1
Tinea infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 6
Blood albumin decreased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 6
Blood amylase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 3
Blood creatinine increased (Investigations) | 1
Blood glucose increased (Investigations) | 5
Blood thyroid stimulating hormone decreased (Investigations) | 4
Blood thyroid stimulating hormone increased (Investigations) | 9
Blood urea increased (Investigations) | 1
Blood urine present (Investigations) | 7
Haemoglobin decreased (Investigations) | 1
Lipase increased (Investigations) | 5
Platelet count decreased (Investigations) | 5
Thyroxine free decreased (Investigations) | 1
Thyroxine free increased (Investigations) | 3
Tri-iodothyronine free increased (Investigations) | 3
Urine bilirubin increased (Investigations) | 2
Weight decreased (Investigations) | 4
White blood cell count decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Lacunar infarction (Nervous system disorders) | 1
Post herpetic neuralgia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 2
Proteinuria (Renal and urinary disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.